CLINICAL TRIAL: NCT03498937
Title: Effet de la tDCS Sur l'impulsivité Chez Les Personnes Souffrant d'un Trouble Borderline : TIMBER
Brief Title: Effects of tDCS on Impulsiveness Among People Suffering From Borderline Personality Disorder
Acronym: TIMBER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P/2017/319
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-04

CONDITIONS: Borderline Personality Disorder; Impulsive Behavior
Keywords: Borderline Personality Disorder; Impulsive behavior; Suicidal behavior; Cognitive control; tDCS; Noninvasive brain stimulation
MeSH Terms: conditions — Borderline Personality Disorder; Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Subjects suffering from Borderline Personality Disorder randomly assigned to start the trial by 10 active tDCS sessions, followed by 10 sham tDCS sessions
  Interventions: Device: Active tDCS; Device: Sham tDCS
- Group 2 (Experimental): Subjects suffering from Borderline Personality Disorder randomly assigned to start the trial by 10 sham tDCS sessions, followed by 10 active tDCS sessions
  Interventions: Device: Active tDCS; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — 10 active tDCS sessions (2 sessions/day for 5 days, 30 min each, 2 mA) applied to the dlPFC
  Other Names: Starstim® (Neuroelectrics, Spain)
Device: Sham tDCS — 10 sham tDCS sessions (2 sessions/day for 5 days, 30 min each, 0 mA) applied to the dlPFC
  Other Names: Starstim® (Neuroelectrics, Spain)

SUMMARY:
The study aims to evaluate the impact of transcranial direct current stimulation (tDCS) on impulsiveness of adults suffering from Borderline Personality Disorder. Short- and long-term effects are assessed by electroencephalography (EEG) records, experimental tasks and self-rated scales.

DETAILED DESCRIPTION:
Impulsivity, considered as the tendency to express spontaneous, excessive and/or unplanned behavior, is recognized as a major factor involved in suicidal behavior and self-harm behaviors. It consists in one of the diagnostic criteria of Borderline Personality Disorder, allowing as well assessment of its clinical severity. There is so far no specific treatment concerning impulsivity. From a neurobiological perspective, the prefrontal cortex is considered as a critical region in the cognitive control of behaviors. Previous studies have associated an hypoactivation of the dorsolateral prefrontal cortex (dlPFC) and the dorsal part of the anterior cingulate cortex to Borderline Personality Disorder.

Transcranial direct current stimulation (tDCS) is a technique of noninvasive brain stimulation which delivers a subthreshold electrical current to the scalp, manipulating the resting membrane potential. It has shown cognitive function improvement, both in healthy individuals and psychiatric populations. Modulation of the dlPFC could therefore represent a mean of reducing impulsivity in those patients.

With a prospective, sham-controlled, crossover, double-blind design, this study aims to evaluate the impact of bilateral tDCS over the dlPFC on the impulsive dimension of adults suffering from Borderline Personality Disorder. Subjects will be submitted to 10 tDCS stimulation sessions (active or sham) for five consecutive days (2 sessions of 30 minutes/day). Current intensity will be of 2 mA, through 25 cm² surface electrodes, placed over the dlPFC (anode position over F4 and cathode over F3, according to the EEG 10-20 international system). Subjects who undergo active stimulation sessions will be then submitted to sham sessions and vice-versa. Baseline measures will be compared to those obtained immediately after the end of sessions (5 days: short-term effects), and to 12 and 30 days later (long-term effects). Active and sham stimulation sessions outcomes will as well be compared.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman older than 18 years old
* Right-handed
* Signed Informed Consent form
* Subject affiliated to or beneficiary from a French social security regime
* Inpatient or outpatient at the Adult Psychiatry Service
* Diagnosis of Borderline Personality Disorder according to the 5th edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria and confirmation by the Structured Clinical Interview for DSM Disorders (SCID-II)
* Absence of addictive comorbidities (except: tobacco, tea, coffee)
* Absence of severe progressive neurologic and/or somatic pathologies (specially tumors, degenerative diseases)

Exclusion Criteria:

* Younger than 18 years old
* Left-handed
* Subject under measure of protection or guardianship of justice
* Presence of psychiatric comorbidities (chronic psychosis, Bipolar Disorder)
* Subject beneficiary from a legal protection regime
* Subject unlikely to cooperate or low cooperation stated by investigator
* Subject not covered by social security
* Pregnant woman
* Subject being in the exclusion period of another study or provided for by the "National Volunteer File"

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
EPs during BART | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Amplitude variation of evoked potentials (EPs) detected by electroencephalography (EEG) during the Balloon Analogue Risk Task (BART), assessing risk-taking behavior. Variation will be obtained by comparing records before beginning of stimulation sessions with 5, 12 and 30 days after active and/or sham tDCS.

SECONDARY OUTCOMES:
BIS-10 scores | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Compared scores from the French version of the Barratt Impulsiveness Scale (BIS-10). The French version of the BIS-10 is a self-rated 34 item questionnaire, composed by three subscales: motor-impulsivity, cognitive-impulsivity and non-planning-impulsivity. Each item is scored on a 0 to 4 points scale. Higher scores indicate higher levels of impulsivity.
HDRS scores | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Compared scores from the Hamilton Depression Rating Scale (HDRS). The HDRS is a clinician-rated 17 item scale which allows depression severity assessment and follow-up. Each item is scored on a 3 or 5 point scale. Scores are represented as follows: 0-7 Normal, 8-13 Mild Depression, 14-18 Moderate Depression, 19-22 Severe Depression, ≥23 Very Severe Depression.
UPPS-P scores | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Compared scores from the Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency Impulsive Behavior Scale (UPPS-P). The French version of the UPPS-P is a self-rated 45 item scale, evaluating the following components: urgency, lack of premeditation, lack of perseverance and sensation seeking. Each item is scored on a base of 4 points. Higher scores indicate higher levels of impulsivity.
MADRS scores | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Compared scores from the Montgomery and Asberg Depression Rating Scale (MADRS). The MADRS is clinician-rated 10 item scale, scored in a base of 6 points per item. Cutoff points are: 0-6 Asymptomatic, 7-19 Mild Depression, 20-34 Moderate Depression and >34 Severe Depression.
C-SSRS scores | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Compared scores from the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS is a clinician-rated tool that evaluates suicidal ideation and behavior. It is composed by 6 "yes/no" questions. High suicide risk is indicated when "yes" is answered to questions 4, 5 or 6.
Go/No-Go task | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Compared results from the experimental Go/No-Go task, assessing response inhibition.
Stroop task | Baseline (Day 0), Day 5, Day 12 and Day 30 post-tDCS
  Compared results from the experimental Stroop task, assessing response inhibition.

CONTACTS AND LOCATIONS:
Overall Officials: Djamila BENNABI, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (3):
- France (3):
  - CHU Besancon, Besançon, Franche-Comte
  - Pôle Hospitalo-Universitaire de Psychiatrie du Grand Nancy, Nancy
  - Centre Hospitalier Spécialisé de Rouffach, Rouffach

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Teti Mayer J, Nicolier M, Gabriel D, Masse C, Giustiniani J, Compagne C, Vandel P, Pazart L, Haffen E, Bennabi D. Efficacy of transcranial direct current stimulation in reducing impulsivity in borderline personality disorder (TIMBER): study protocol of a randomized controlled clinical trial. Trials. 2019 Jun 10;20(1):347. doi: 10.1186/s13063-019-3427-z. PMID 31182143